CLINICAL TRIAL: NCT00697892
Title: Pharmacokinetic Interactions Between Antiretroviral Agents, Lopinavir/Ritonavir and Efavirenz and Antimalarial Drug Combinations, Artesunate/Amodiaquine and Artemether/Lumefantrine.
Brief Title: Pharmacokinetic Interactions Between Antiretroviral Agents and Antimalarial Drug Combinations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fran Aweeka (Other)
Responsible Party: Sponsor-Investigator, Fran Aweeka, Sponsor-Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H6930-27654
Record Dates: First submitted 2008-06-02; First posted 2008-06-16 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-05

CONDITIONS: HIV Infections; Malaria
Keywords: Human Immunodeficiency Virus; Drug Interactions
MeSH Terms: conditions — HIV Infections; Malaria; Acquired Immunodeficiency Syndrome | interventions — Lopinavir; lopinavir-ritonavir drug combination; efavirenz; Artemether, Lumefantrine Drug Combination

ARMS (2):
- Group A4 (Experimental): healthy volunteers assigned to the efavirenz with artemether/lumefantrine intervention
  Interventions: Drug: efavirenz; Drug: artemether/lumefantrine
- Group A3 (Experimental): healthy volunteers assigned to the lopinavir/ritonavir with artemether/lumefantrine intervention
  Interventions: Drug: lopinavir/ritonavir; Drug: artemether/lumefantrine

INTERVENTIONS:
Drug: lopinavir/ritonavir — Two tablets of lopinavir 200mg / ritonavir 50mg orally twice daily with food for 26 days
  Other Names: Kaletra
  Arms: Group A3
Drug: efavirenz — One 600mg tablet orally once daily before bedtime on an empty stomach for 26 days
  Other Names: Sustiva
  Arms: Group A4
Drug: artemether/lumefantrine — 4 tablets of artemether 20mg/lumefantrine 120mg twice daily with food. 2 three-day courses will be administered (with washout in between) during the duration of the trial.
  Other Names: Coartem

SUMMARY:
The purpose of the study is to determine in healthy volunteers whether certain anti-HIV medications (lopinavir/ritonavir and efavirenz) affect the drug levels of certain anti-malarial medications (artesunate/ amodiaquine and artemether/ lumefantrine) and vice versa. Since these drugs are degraded using overlapping pathways in the liver, it is predicted that changes in both drug level and overall drug exposure will be observed.

DETAILED DESCRIPTION:
HIV and malaria are two of the most pernicious diseases facing developing countries. Malaria affects 300 to 500 million individuals annually in developing countries and it is estimated that 25.8 million people in Africa live with HIV. Current therapy recommended by the World Health Organization includes the use of artemisinin derivatives, such as artesunate and artemether. To minimize the risk of resistance, these drugs are used in combination with older drugs with longer half-lives including amodiaquine and lumefantrine.

Treatment of malaria is further complicated by the increasing availability of antiretroviral (ARV) medications for HIV in that clinically important drug-drug interactions may occur in co-infected patients. Protease inhibitor (e.g. lopinavir and ritonavir) and non-nucleoside reverse transcriptase (e.g. efavirenz) based treatment commonly affects pharmacokinetic exposure of drugs metabolized by cytochrome P450 (CYP) metabolic pathways.

Artemether is metabolized by the CYP3A4 to active dihydroartemisinin (DHA), while artesunate is hydrolyzed to DHA. Lumefantrine is an active compound that is metabolized by CYP3A4. Amodiaquine is an active "prodrug" that is quickly metabolized to an active metabolite N-desethylamodiaquine (DEAQ) by CYP2C8. In addition, these antimalarial drugs may also affect the metabolism of CYP substrates, such as ARVs.

The primary objective of this study is to investigate the effects of ARV agents (ritonavir/ lopinavir (Kaletra) and efavirenz) on the pharmacokinetics of antimalarial drug combinations [artesunate/ amodiaquine and their active metabolites, and artemether/ lumefantrine (Coartem®) and their active metabolites]. The secondary objective is to investigate the effects of antimalarial drug combinations [artesunate/amodiaquine and artemether/lumefantrine (Coartem®)] on the pharmacokinetics of ARV drugs [lopinavir/ritonavir (Kaletra®) and efavirenz].

If clinically important interactions occur, net effects may include improved or diminished antimalarial activity (as activity is attributed to both the parent drug and the active metabolite(s)) and drug toxicity. The study in HIV negative healthy volunteers will allow rapid assessment of these potential interactions and will provide essential data for optimizing a future clinical study and the use of ARVs and antimalarials for children and adults in Uganda.

Currently the components of the study involving the impact of ARVs on artesunate/amodiaquine are not being pursued (and recruitment for those arms was conducted separately), so there are only two groups in the presently-approved trial: one in which the effects of lopinavir/ritonavir on artemether/lumefantrine are studied and another in which the effects of efavirenz on artemether/lumefantrine are studied.

ELIGIBILITY:
Inclusion Criteria:

* Absence of HIV infection prior to study entry
* Male or female aged 21-60 who are able to provide informed consent
* Subject is within 20% (+/-) of ideal body weight and weighs at least 50 kg.
* Healthy, without evidence of acute or chronic illness including diabetes, hypertension, CAD, psychiatric illnesses, renal or hepatic impairment.
* Screening laboratory tests that are normal or deemed not clinically significant by the study physician.
* Female subjects of reproductive potential must agree to the use of two forms of birth control methods for at least one month prior to study enrollment and for 6 weeks following study completion
* Female subjects must have a negative pregnancy test within 24 hours before receiving any study drugs.

Exclusion Criteria:

* Use of illicit drugs or alcohol that could interfere with the completion of the study
* Use of any over-the-counter or prescribed drugs unless approved by the principal investigator or study physician
* Use of drugs that are known to inhibit/induce CYP450 isozymes or are substrates of CYP3A4, CYP2D6, CYP2C8 enzymes (use of hormonal contraceptives is permitted).
* Pregnant or breastfeeding
* History of acute or chronic illnesses, such as diabetes, hypertension, CAD, psychiatric illnesses, renal or hepatic impairment.
* Evidence of acute illness
* Family history of congenital prolongation of QTc interval or with any conditions known to prolong QTc interval such as cardiac arrhythmias, bradycardia, or severe heart disease
* History of hypokalemia, hypomagnesemia, or hypercholesteremia

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2005-07; Primary Completion 2008-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
AUC (zero to infinity) of the antimalarial agent | Each 3-day antimalarial treatment course throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Francesca T Aweeka, PharmD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States